CLINICAL TRIAL: NCT06266039
Title: A Prospective Observational Study in Naturalistic Settings to Describe Long Acting Buprenorphine Introduction in France: Change in Severity of Addiction and Health Related Quality of Life Over a Period of 6 Months.
Brief Title: Introduction of Long Acting Buprenorphine in France
Acronym: OBAP
Status: Recruiting | Type: Observational
Sponsor: University of Bordeaux (Other)
Responsible Party: Principal Investigator, Marc Auriacombe, Professor, University of Bordeaux
Other Study IDs: 2022-0328-01; 2022-A02616-37 (Other: French National Agency for the Safety of Medicines (ANSM))
Record Dates: First submitted 2023-08-28; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Addiction Opiate
Keywords: opioid use disorder (OUD); patient reported outcome measure (PROM); addiction severity index (ASI); long acting buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
The current available pharmacological treatment formulations (i.e., daily formulations of buprenorphine or methadone) for OUD in France may have several inconveniences, such as: compliance, burden of daily intake, and risk of misuse; that may hinder their effectiveness. Long acting formulations of buprenorphine (LAB) such as Buvidal have been developed to favor retention and compliance and minimize the risk of diversion. Previous studies are promising on the advantage of LAB to treat opioid addiction, however more evidence is needed in the French healthcare context. However, in addition to randomized clinical trials, the French National Healthcare Agency (HAS "Haute Autorité de Santé") recommends conducting "real-life" studies (i.e., in naturalistic conditions) during the development of a medication and the use of "Patient Reported Outcome Measures" (PROMs) to analyze patient quality of life and/or other measures relevant to patients (e.g., severity, efficiency), without interpretation of the answers by a health professional. In this regard, our study proposes to use the Addiction Severity Index (ASI) self-report questions and several scales on treatment satisfaction and quality of life to collect the patient's opinion of perceived changes following the use of Buvidal.

Main objectives:

The objectives of this prospective open observational study, in naturalistic conditions, are to examine in individuals with an opioid use disorder, over a period of 6 months after LAB treatment initiation: the change in substance addiction severity and the changes in health-related quality of life, craving, opioids and other substance and non-substance uses and misuses, alcohol, tobacco and non-substance addiction severity, satisfaction with LAB treatment, severity of others domains related to addiction severity (i.e., medical, social, psychological) and psychiatric comorbidities

Main hypotheses:

1. Hypothesize was that LAB will be associated with a stable (if prior remission) or a reduction of the CS of "Drug use" (i.e., substance addiction severity) at 6 months compared to baseline.
2. Hypothesize was that LAB will be associated with a stable (if prior remission) or a reduction of opioids and other substance and non-substance uses and misuses, other substances and non-substances addiction severity, craving, severity of others domains related to addiction (i.e., medical status, employment and support, family/social status, psychological status), an improvement of quality of life and a good satisfaction with treatment at follow-ups compared to baseline.

DETAILED DESCRIPTION:
Context The current available pharmacological treatment formulations (i.e., daily formulations of buprenorphine or methadone) for OUD in France may have several inconveniences, such as: compliance, burden of daily intake, and risk of misuse; that may hinder their effectiveness. Long acting formulations of buprenorphine (LAB) such as Buvidal have been developed to favor retention and compliance and minimize the risk of diversion. The previous studies are promising on the advantage of LAB to treat opioid addiction, however more evidence is needed in the French healthcare context.

In a French pilot study of Buvidal initiation, one third of subjects stopped Buvidal treatment prematurely (before the 3-month follow-up) but some were back on treatment at the 6-month follow-up. Buvidal seems to be promising to maintain patients in treatment, compared to daily buprenorphine, but there are late drop-outs and some of the early drop-outs may resume treatment. A 6 months follow-up would allow to explore this phenomenon and better characterize medium term LAB compliance.

None of the previous or underway studies examined the effect of Buvidal on craving over time or the cues-craving-use relationship in daily life. Chronic opioid use generates intense reactivity to opioid-conditioned cues, including craving and opioid seeking behavior. Craving is a very dynamic phenomenon across a day and its variations are best captured by Ecological Momentary Assessment (EMA) method. Previous EMA studies from SANPSY highlighted a unidirectional prospective link between cues, craving and use. EMA method would be appropriate to describe the effect of Buvidal on craving, opioid use, and the relationship between cues, craving and opioid use.

In addition to randomized clinical trials, the French National Healthcare Agency (HAS "Haute Autorité de Santé") recommends conducting "real-life" studies (i.e., in naturalistic conditions) during the development of a medication and the use of "Patient Reported Outcome Measures" (PROMs) to analyze patient quality of life and/or other measures relevant to patients (e.g., severity, efficiency), without interpretation of the answers by a health professional. However, the absence of a control group could overlook several important potential biases. In the context of this study, a randomized control trial (RCT) design would not be appropriate, but the use of a Historical Cohort control group design is an alternative. ADDICTAQUI is an ongoing longitudinal naturalistic open cohort ongoing since 1994 at SANPSY/University of Bordeaux. It includes participants initiating treatment for OUD and uses assessments similar to the current study.

In this regard, our study proposes to use the Addiction Severity Index (ASI) self-report questions and several scales on treatment satisfaction and quality of life to collect the patient's opinion of perceived changes following the use of Buvidal.

Objectives

The objectives of this prospective open observational study, in naturalistic conditions, are to examine in individuals with an opioid use disorder, over a period of 6 months after LAB treatment initiation:

1. the change in substance addiction severity
2. the changes in health-related quality of life, craving, opioids and other substance and non-substance uses and misuses, alcohol, tobacco and non-substance addiction severity, satisfaction with LAB treatment, severity of others domains related to addiction severity (i.e., medical, social, psychological) and psychiatric comorbidities
3. to compare craving intensity reported in daily life, and mood, insight, self-efficacy, cues, opioid use, other substances and non-substance use, and the links between cues and craving, and between craving and opioid use, in daily life before and after LAB initiation within subjects
4. to compare the 6-month outcomes of individuals initiating LAB treatment to an historical control group of individuals initiating daily buprenorphine or methadone within the ADDICTAQUI Cohort
5. to explore factors associated to dropout of LAB treatment at 6-month follow-ups and factors associated to resuming LAB at 6 months after previous drop-out

Evaluation criteria

* Main: Composite score of the "Drug use" section from the ASI.
* Secondary: Quality of life (EQ-5D-5L, NHP, SF-12, ASI, TEAQV), addiction severity (ASI, MINI), opioid use and misuse (ASI), others substance and non-substance use and misuse (ASI), alcohol, tobacco and non-substance addiction severity (ASI), craving (Craving Scale), severity of other domains related to addiction (i.e., medical, social, professional, familial, psychological (ASI)), treatment satisfaction (TSQM), socio-demographic characteristics (ASI), psychiatric comorbidities (MINI), treatment history (ASI) and acceptability and acceptance of treatment by prescribing physician.

Hypotheses

1. Hypothesize was that LAB will be associated with a stable (if prior remission) or a reduction of the CS of "Drug use" (i.e., substance addiction severity) at 6 months compared to baseline.
2. Hypothesize was that LAB will be associated with a stable (if prior remission) or a reduction of opioids and other substance and non-substance uses and misuses, other substances and non-substances addiction severity, craving, severity of others domains related to addiction (i.e., medical status, employment and support, family/social status, psychological status), an improvement of quality of life and a good satisfaction with treatment at follow-ups compared to baseline.
3. Hypothesize was that LAB will be associated with a stable (if prior remission) or a reduction of craving (intensity/frequency), opioid use and other substances and non-substance-uses, and an improvement of mood, insight, self-efficacy. We also hypothesize that LAB will be associated with a reduction in the association between cues and craving, and the association between craving and opioid use, in daily life.
4. Hypothesize was that LAB group would have better outcomes after 6 months of treatment compared to the historical control group: with lower severity of addiction, higher quality of life and treatment adherence among patients with OUD, when controlling for baseline characteristics (e.g., socio-demographics factors and addiction severity).
5. Exploratory analyses will be conducted to assess what are the predictors of LAB treatment adherence at 6 months.

Benefit/Risk Balance This observational study has a favorable benefit/risk ratio for all participants.

Study design This study is a 6 months prospective open observational study in naturalistic conditions, recruiting patients (n=223) initiating LAB treatment in French Addiction Treatment Centers (i.e., Centre de Soins, d'Accompagnement et de Prévention en Addictologie (CSAPA), services hospitaliers d'addictologie) or in French penitentiary centers, which are currently the only way to access LAB (Buvidal).

All participants will receive a baseline assessment before LAB initiation, 4 follow-up assessments at 1, 2, 3 and 6 months after treatment initiation.

All evaluations will be conducted by phone by Clinical Research Assistants (CRAs) and online questionnaires. CRAs of University of Bordeaux, SANPSY lab, that do not take part in the interventions, will be trained in research evaluations, including the collection of standardized data by phone using reliable and efficient evaluation tools. A procedure will be put in place to ensure perfect homogeneity among all evaluators involved in the study.

A sub-sample of participants (n=68) will also receive 4 weeks of EMA procedure using an app downloaded on participant's smartphone.

ELIGIBILITY:
Inclusion Criteria:

* To have been prescribed LAB
* To plan to initiate a LAB treatment in the following month
* To be over 18 years of age
* To accept to participate after an informed consent procedure

Exclusion Criteria:

* To be under guardianship, curatorship or safeguard of justice
* To have a difficulty understand / reading the French language
* To have any condition incompatible with study participation (e.g., not being able to communicate by phone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants included in this observational study in the French healthcare context will be recruited from the current prescribers of LAB, which are medical doctors working in Addiction Treatment Centers (i.e., Centre de Soins, d'Accompagnement et de Prévention en Addictologie (CSAPA), services hospitaliers d'addictologie) in France.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The change in the composite score of the "Drug use" section from the Addiction Severity Index (ASI) at 6 months after treatment initiation | At 6 months compared to baseline
  The main outcome criteria will be the change in substance addiction severity (i.e., composite score of "Drug section" of the ASI which is a standard multidimensional measure, range from 0 "no drug problem" to 1 "extreme drug problem") during the first 6 months of LAB treatment initiation in individuals with an opioid use disorder, in the French health care context.

SECONDARY OUTCOMES:
The change in addiction severity at 6 months after treatment initiation | At 6 months compared to baseline
  Addiction Severity Index (ASI): trouble and treatment need in the past 30 days; from 0=not at all to 4=extremely
The change in quality of life with EuroQoL-5 Dimensions-5 Levels (EQ-5DL-5L) at 6 months after treatment initiation | At 6 months compared to baseline
  EQ-5D-5L describes five dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Respondents are asked to choose the statement in each dimension that best describes their health status on the day they are surveyed. Their responses are coded as a number (1 to 5) that corresponds to the respective level of severity.
The change in quality of life with the 12-Item Short Form Survey (SF-12) at 6 months after treatment initiation | At 6 months compared to baseline
  SF-12: physical and emotional component scores (0-100 points). Higher score indicates a better health.
The change in quality of life with nottingham health profile part 1 and part 2 (NHP1 and NHP2) at 6 months after treatment initiation | At 6 months compared to baseline
  NHP1/ NHP2: 45 items (yes/no each coded as 1/0). Items in each domain are assigned a weight; the total score for each domain is 100 points where a score of 0 indicates good subjective health status and 100 indicates poor subjective health status. The NHP total score is obtained by averaging the six domain scores. Higher score indicates a greater perceived distress in each dimension.
The change in quality of life with assisted quality of life assessment chart (TEAQV) at 6 months after treatment initiation | At 6 months compared to baseline
  TEAQV: 7 point-scale (0=extremely bad; 6=excellent) according 4 dimensions: physical and psychological well-being, family relationships, professional activity
The change in other use at 6 months after treatment initiation | At 6 months compared to baseline
  Other uses: number of days of use (0-30 days) and number of intakes per day, Composite Scores of the Addiction Severity Index ranging from 0 to 1.
The change in craving at 6 months after treatment initiation | At 6 months compared to baseline
  Craving: number of days (0-30 days), craving mean and maximal intensities (0=no craving to 10=extreme craving)
The change in other domains of addiction severity at 6 months after treatment initiation | At 6 months compared to baseline
  Severity of others domains: medical, employment and support, family/social, psychological; Composite Scores (from 0 no problem to 1 extreme problem)
The change in Treatment Satisfaction Questionnaire for Medication (TSQM) at 6 months after treatment initiation | At 6 months compared to baseline
  TSQM: effectiveness, side effects, convenience, and global satisfaction; from 0 to 100 points, with a higher score indicating a better satisfaction
Cues - craving - use links and others factors variations measure with EMA after treatment initiation | From 1 to 14 days after treatment initiation
  Use of EMA data to compare craving intensity,mood, insight, self-efficacy, cues, opioids use, other substances and non-substance use, and the links between cues and craving, and between craving and opioid use, in daily life before and after LAB initiation
  * Anxiety (1 = no anxiety to 7 = extreme anxietey)
  * Sadness (1 = no sadness to 7 = extreme sadness)
  * Happiness ((1 = no happiness to 7 = extreme happiness)
  * Insight (1 = low insight to 7 = high insight)
  * Self-efficacy (1 = no self-efficacy to 7 = excelletent self-efficacy)
  * Number of cues
  * Intensity of craving (1 = no craving to 7 = extreme craving)
  * Opioids use (0 = no ; 1 = yes)
  * Other substances and non-substances use (0 = no ; 1 = yes)
  * Prospective association between number of cues and craving intensity (coefficient of correlation between cues and craving)
  * Prospective association between craving intensity and substance use (coefficient of correlation between craving and use)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bordeaux, Bordeaux, Gironde, France